CLINICAL TRIAL: NCT03392727
Title: Evaluation of Safe Sleep for Babies: a Bassinet Distribution and Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Paediatric Society (Other); Manitoba Health, Seniors and Active Living (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2017:390
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-01

CONDITIONS: Sudden Infant Death
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Box & Education Session (Experimental): Parents are provided a baby box and infant health and safety products and participate in a face to face educational session
  Interventions: Device: Study Box; Behavioral: Education Session
- Community Box & Online Education (Active Comparator): Parents are informed how to receive a free box from a community site and are provided a guide to online resources for prenatal and infant health promotion
  Interventions: Device: Community Box; Behavioral: Online Education

INTERVENTIONS:
Device: Study Box — Baby box (bassinet) with infant items
  Arms: Study Box & Education Session
Device: Community Box — Baby box (bassinet)
  Arms: Community Box & Online Education
Behavioral: Education Session — Face to face education and baby box orientation session
  Arms: Study Box & Education Session
Behavioral: Online Education — Online baby box education
  Arms: Community Box & Online Education

SUMMARY:
This study will evaluate baby box ownership and safe sleep practices (sleep location, sleep position, use of bedding) among families provided a free baby box and standardized safe sleep education compared to families provided a safe sleep pamphlet and information on how to obtain a free box in the community.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial with two arms: the intervention group (n=110) will be provided a baby box and standardized face to face education regarding the box and its contents, safe sleep, and infant health promotion; the control group (n=110) will be provided information on how to obtain the same baby box at a community site in Winnipeg, and will receive a safe sleep pamphlet, baby box pamphlet and a guide to online resources for prenatal ad infant health promotion. An additional comparison group will be parents who already have a baby box at the time of recruitment. This group will also receive the safe sleep pamphlet. Families will be interviewed at recruitment and 2-4 months of age to measure box ownership and self-reported safe sleep and infant health promotion practices. Administrative data will be used to evaluate the impact on infant immunizations and hospitalizations in the first year of life, and to evaluate the impacts of prenatal care visits and neonatal length of stay on the outcomes.

Families will be asked to participate in a face to face interview at baseline (enrolment) and one follow-up interview coordinated with a scheduled routine healthcare visit for the infant at 2 months of age and conducted face to face or by telephone, according to family preference.

PHIN will be requested for both mother and infant in order to explore the relationship between adequacy of prenatal care and the study outcomes, and to evaluate the impact on infant immunizations and hospitalizations in the first year of life. Postal code will be requested to analyze differences related to place of residence and neighbourhood income quintile.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are 32 weeks or more gestation
* Infants less than 3 months of age (or post-conceptional age 44 weeks)
* Able to consent freely and complete face to face and/or telephone interviews in English
* Will be residing in Winnipeg until the infant is 2-4 months of age or able to complete a telephone interview at 2-4 months of age

Exclusion Criteria:

* Parent/guardian/client less than 18 years of age (unless emancipated minor)
* Parents who cannot consent due to intellectual capacity, medical condition, etc.
* Infant is discharged from hospital in the care of Child and Family Services or a birth alert is in place

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Box ownership | 2 months
  Parents with a baby box
Usual sleep location | 2 months
  crib, cradle, bassinet, box, other
Baby box use for sleep | 2 months
  always/sometimes/never/not applicable
Usual sleep position | 2 months
  supine, other
Usual infant clothing for sleep | 2 months
  sleeper, sack, swaddled
Usual bedding | 2 months
  none, tucked blanket, other

SECONDARY OUTCOMES:
Safe sleep knowledge | 2 months
  safe sleep location, position, infant clothing, bedding (1 point each)
Current infant feeding | 2 months
  breastfeeding, formula feeding, both
Household smoking | 2 months
  total number of cigarettes smoked per day in the household
Vitamin D | 2 months
  Infant provided daily dose of Vitamin D (always/sometimes/never)
Immunizations | 12 months
  Number of infant immunizations in the first year of life
Prenatal visits | 9 months
  Number of prenatal visits
Infant hospitalizations | 12 months
  Infant hospitalizations in the first year of life (number of hospitalizations, total hospital days, respiratory vs. non-respiratory hospital days)

OTHER OUTCOMES:
Adverse events | 2 months
  Parent-reported adverse events and concerns regarding the baby box
Parent feedback | 2 months
  Parent-reported opinions and preferences (likes/dislikes) regarding the baby box and the distribution process

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Nickel, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No